CLINICAL TRIAL: NCT02728596
Title: A Pragmatic Trial to Evaluate a Guideline-Based Colony Stimulating Factor Standing Order Intervention and to Determine the Effectiveness of Colony Stimulating Factor Use as a Prophylaxis for Patients Receiving Chemotherapy With Intermediate Risk for Febrile Neutropenia - Trial Assessing CSF Prescribing Effectiveness and Risk (TrACER)
Brief Title: S1415CD, Trial Assessing CSF Prescribing Effectiveness and Risk (TrACER)
Acronym: TrACER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: S1415CD; NCI-2016-00264 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1415; S1415CD (Other: SWOG); SWOG-S1415CD (Other: DCP); UG1CA189974 (NIH)
Record Dates: First submitted 2016-03-30; First posted 2016-04-05 (Estimated); Results first posted 2022-10-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-09

CONDITIONS: Febrile Neutropenia; Stage 0 Breast Cancer; Stage 0 Colorectal Cancer; Stage 0 Non-Small Cell Lung Cancer; Stage I Colorectal Cancer; Stage IA Breast Cancer; Stage IA Non-Small Cell Lung Carcinoma; Stage IB Breast Cancer; Stage IB Non-Small Cell Lung Carcinoma; Stage IIA Breast Cancer; Stage IIA Colorectal Cancer; Stage IIA Non-Small Cell Lung Carcinoma; Stage IIB Breast Cancer; Stage IIB Colorectal Cancer; Stage IIB Non-Small Cell Lung Carcinoma; Stage IIC Colorectal Cancer; Stage IIIA Breast Cancer; Stage IIIA Colorectal Cancer; Stage IIIA Non-Small Cell Lung Cancer; Stage IIIB Breast Cancer; Stage IIIB Colorectal Cancer; Stage IIIB Non-Small Cell Lung Cancer; Stage IIIC Breast Cancer; Stage IIIC Colorectal Cancer; Stage IV Breast Cancer; Stage IV Non-Small Cell Lung Cancer; Stage IVA Colorectal Cancer; Stage IVB Colorectal Cancer
MeSH Terms: conditions — Febrile Neutropenia; Breast Carcinoma In Situ; Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Clinic group 1 (clinics with existing automated system for CSF prescribing) (Active Comparator): CSF prescribing for patients taking anti-cancer drugs is based on existing automated system recommendations: CSF is recommended for drugs with high risk of FN; CSF is not recommended for drugs with low risk of FN.
  Interventions: Other: Preventive Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Clinic group 2 (clinics with no automated system for CSF prescribing) (Active Comparator): CSF prescribing for patients taking anti-cancer drugs is based on existing clinical practice guidelines.
  Interventions: Other: Preventive Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Clinic group 3 (clinics with automated system for CSF prescribing) (Experimental): CSF prescribing for patients taking anti-cancer drugs is based on automated system recommendations: CSF is recommended for drugs with intermediate or high risk of FN; CSF is not recommended for drugs with low risk of FN.
  Interventions: Other: Preventive Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Clinic group 4 (clinics with automated system for CSF prescribing) (Experimental): CSF prescribing for patients taking anti-cancer drugs is based on automated system recommendations: CSF is recommended for drug with high risk of FN; CSF is not recommended for drugs with intermediate or low risk of FN.
  Interventions: Other: Preventive Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Preventive Intervention — Automated ordering system recommends prescribing or not prescribing CSF based on drug's risk level for FN
  Other Names: PREVENTATIVE; Prevention; Prevention Measures; Prophylaxis; PRYLX
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized clinical trial studies prophylactic colony stimulating factor management in patients with breast, colorectal or non-small cell lung cancer receiving chemotherapy and with risk of developing febrile neutropenia. Patients receiving chemotherapy may develop febrile neutropenia. Febrile neutropenia is a condition that involves fever and a low number of neutrophils (a type of white blood cell) in the blood. Febrile neutropenia increases the risk of infection. Colony stimulating factors are medications sometimes given to patients receiving chemotherapy to prevent febrile neutropenia. Colony stimulating factors are given to patients based on guidelines. Some clinics have an automated system that helps doctors decide when to prescribe them when there is a high risk of developing febrile neutropenia. Gathering information about the use of an automated system to prescribe prophylactic colony stimulating factor may help doctors use colony stimulating factor when it is needed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the use of primary prophylactic colony stimulating factor (PP-CSF) according to recommended clinical practice guidelines among patients registered at intervention components versus usual care components.

II. To compare the rate of febrile neutropenia (FN) among patients registered at intervention components versus usual care components.

III. To compare the rate of FN among intermediate risk patients registered at intervention components by component treatment assignment (administer PP-CSF to intermediate risk patients versus not).

SECONDARY OBJECTIVES:

I. To compare the rate of FN among low-risk patients registered at intervention components versus usual care components.

II. To compare the FN-related health-related quality of life (HRQOL) among low-risk patients registered at intervention components versus usual care components.

III. To compare patient adherence to PP-CSF prescribing among patients registered at intervention components versus usual care components.

IV. To compare patient knowledge of the indications for, efficacy of, and side effects associated with PP-CSF between the initiation and conclusion of the first cycle of myelosuppressive systemic therapy among patients registered at intervention components versus usual care components.

V. To compare the proportion of patients completing the initial systemic therapy regimen at planned duration and at planned dose intensity among patients registered at intervention components versus usual care components.

VI. To compare antibiotic use both as prophylaxis and as treatment for FN among patients registered at intervention components versus usual care components.

VII. To compare the rate of FN-related emergency department visits and hospitalizations among intermediate risk patients registered to Intervention components by component treatment assignment (administer PP-CSF to intermediate risk patients versus not).

VIII. To compare the FN-related health-related quality of life (HRQOL) among intermediate risk patients registered to intervention components by component treatment assignment (administer PP-CSF to intermediate risk patients versus not).

IX. To compare overall survival among intermediate risk patients registered to intervention components by component treatment assignment (administer PP-CSF to intermediate risk patients versus not).

TERTIARY OBJECTIVES:

I. To characterize and descriptively report the differences among cohort components and the intervention and usual care components.

II. To evaluate the time to invasive recurrence in non-metastatic patients by component treatment assignment

OUTLINE: Patients are randomized to 1 of 4 clinic groups.

CLINIC GROUP 1 (CLINIC WITH AUTOMATED SYSTEM): Patients with a high risk of developing FN receive CSF based on the automated system recommendations. The automated system suggests that CSFs not be used for drugs that have a low risk of FN.

CLINIC GROUP 2 (CLINIC WITH NO AUTOMATED SYSTEM): Patients receive CSF based on clinical practice guidelines.

CLINIC GROUP 3 (CLINIC WITH AUTOMATED SYSTEM): Patients with a high or moderate risk of developing FN receive CSF based on the automated system recommendations. The automated system suggests that CSFs not be used for drugs that have a low risk of FN.

CLINIC GROUP 4 (CLINIC WITH AUTOMATED SYSTEM): Patients with a high risk of developing FN receive CSF based on the automated system recommendations. The automated system suggests that CSF not be used for drugs that have a moderate risk of FN.

After completion of study treatment, patients are followed up for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a current diagnosis of breast cancer, non-small cell lung cancer, or colorectal cancer; the current diagnosis may be an initial diagnosis or recurrence and/or progression of previously diagnosed disease; cancer may be metastatic or non-metastatic
* Patients must be registered prior to or on the same day as their first cycle of chemotherapy for their current disease and stage 9or disease setting).
* Patients must not have had any systemic therapy (chemotherapy or combination regimens) in the 180 days just prior to registration. Prior biologic therapy, immunotherapy, tyrosine kinase inhibitors, and hormonal therapy are allowed.
* Patients must be planning to receive one of the study-allowed regimens as their initial treatment for their current disease; myelosuppressive therapy must follow the standard regimen, although a dose reduction of up to 10% is permitted. This treatment may be neoadjuvant or adjuvant chemotherapy.
* Patients must not be receiving or planning to receive concurrent radiation during systemic treatment.
* Patients must not have any known contraindication to CSFs prior to registration, including prior hypersensitivity to Escherichia coli-derived proteins, filgrastim, pegfilgrastim, or tbo-filgrastim
* Patients must be able to understand and provide information for the patient-completed study forms in either English or Spanish
* Patients may have had a prior malignancy
* Patients must not be participating or plan to participate in other clinical trials that involve investigational systemic cancer treatments or investigational uses of CSF during their first 6 months after registration
* Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3665 (Actual)
Dates: Start 2016-10-07 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Ramsey, Principal Investigator — SWOG Cancer Research Network
Locations (160):
- United States (159):
  - Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - NEA Baptist Memorial Hospital, Jonesboro, Arkansas
  - Contra Costa Regional Medical Center, Martinez, California
  - Augusta University Medical Center, Augusta, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute - Nampa, Nampa, Idaho
  - Saint Luke's Mountain States Tumor Institute-Twin Falls, Twin Falls, Idaho
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Cancer Care Specialists of Illinois-Swansea, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center Shreveport, Shreveport, Louisiana
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Presbyterian Rust Medical Center/Jorgensen Cancer Center, Rio Rancho, New Mexico
  - Christus Saint Vincent Regional Cancer Center, Santa Fe, New Mexico
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Novant Health Oncology Specialists-Kernersville, Kernersville, North Carolina
  - Novant Health Oncology Specialists-Mount Airy, Mount Airy, North Carolina
  - Novant Health Oncology Specialists-Statesville, Statesville, North Carolina
  - Novant Health Oncology Specialists-Davidson County, Thomasville, North Carolina
  - Novant Health Oncology Specialists-Wilkesboro, Wilkesboro, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Novant Health Oncology Specialists, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Dayton Physician LLC-Miami Valley Hospital North, Dayton, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Dayton Physicians LLC-Signal Point, Middletown, Ohio
  - Dayton Physicians LLC-Wilson, Sidney, Ohio
  - Dayton Physicians LLC-Upper Valley, Troy, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - MGC Hematology Oncology-Union, Union, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Integrity Oncology PLLC-Collierville, Collierville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Family Cancer Center-Memphis, Memphis, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Marshfield Clinic - Ladysmith Center, Ladysmith, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
- Doctors Cancer Center, Manatí, Puerto Rico

REFERENCES:
- [Derived] Hershman DL, Bansal A, Barlow WE, Arnold KB, Watabayashi K, Bell-Brown A, Sullivan SD, Lyman GH, Ramsey SD. Intervention Nonadherence in the TrACER (S1415CD) Study: A Pragmatic Randomized Trial of a Standardized Order Entry for CSF Prescribing. JCO Oncol Pract. 2023 Dec;19(12):1160-1167. doi: 10.1200/OP.23.00219. Epub 2023 Oct 3. PMID 37788414
- [Derived] Lyman GH, Bansal A, Sullivan SD, Arnold KB, Barlow WE, Hershman DL, Lad TE, Ramsey SD. Impact of treatment experience on patient knowledge of colony-stimulating factors among patients receiving cancer chemotherapy: evidence from S1415CD-a large pragmatic trial. Support Care Cancer. 2023 Sep 28;31(10):598. doi: 10.1007/s00520-023-08056-z. PMID 37770704
- [Derived] Ramsey SD, Bansal A, Sullivan SD, Lyman GH, Barlow WE, Arnold KB, Watabayashi K, Bell-Brown A, Kreizenbeck K, Le-Lindqwister NA, Dul CL, Brown-Glaberman UA, Behrens RJ, Vogel V, Alluri N, Hershman DL. Effects of a Guideline-Informed Clinical Decision Support System Intervention to Improve Colony-Stimulating Factor Prescribing: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2022 Oct 3;5(10):e2238191. doi: 10.1001/jamanetworkopen.2022.38191. PMID 36279134
- [Derived] Hershman DL, Bansal A, Sullivan SD, Barlow WE, Arnold KB, Watabayashi K, Bell-Brown A, Le-Lindqwister NA, Dul CL, Brown-Glaberman UA, Behrens RJ, Vogel V, Alluri N, Ramsey SD. A Pragmatic Cluster-Randomized Trial of a Standing Order Entry Intervention for Colony-Stimulating Factor Use Among Patients at Intermediate Risk for Febrile Neutropenia. J Clin Oncol. 2023 Jan 20;41(3):590-598. doi: 10.1200/JCO.22.01258. Epub 2022 Oct 13. PMID 36228177
- [Derived] Watabayashi KK, Bell-Brown A, Kreizenbeck K, Egan K, Lyman GH, Hershman DL, Arnold KB, Bansal A, Barlow WE, Sullivan SD, Ramsey SD. Successes and challenges of implementing a cancer care delivery intervention in community oncology practices: lessons learned from SWOG S1415CD. BMC Health Serv Res. 2022 Apr 1;22(1):432. doi: 10.1186/s12913-022-07835-4. PMID 35365139

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Comparator: Clinic Group 1 (Clinics With Existing Automated System for CSF Prescribing): CSF prescribing for patients taking anti-cancer drugs is based on existing automated system recommendations: CSF is recommended for drugs with high risk of FN; CSF is not recommended for drugs with low risk of FN.
  Preventive Intervention: Automated ordering system recommends prescribing or not prescribing CSF based on drug's risk level for FN
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
- Active Comparator: Clinic Group 2 (Clinics With no Automated System for CSF Prescribing): CSF prescribing for patients taking anti-cancer drugs is based on existing clinical practice guidelines.
  Preventive Intervention: Automated ordering system recommends prescribing or not prescribing CSF based on drug's risk level for FN
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
- Experimental: Clinic Group 3 (Clinics With Automated System for CSF Prescribing): CSF prescribing for patients taking anti-cancer drugs is based on automated system recommendations: CSF is recommended for drugs with intermediate or high risk of FN; CSF is not recommended for drugs with low risk of FN.
  Preventive Intervention: Automated ordering system recommends prescribing or not prescribing CSF based on drug's risk level for FN
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
- Experimental: Clinic Group 4 (Clinics With Automated System for CSF Prescribing): CSF prescribing for patients taking anti-cancer drugs is based on automated system recommendations: CSF is recommended for drug with high risk of FN; CSF is not recommended for drugs with intermediate or low risk of FN.
  Preventive Intervention: Automated ordering system recommends prescribing or not prescribing CSF based on drug's risk level for FN
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
Period: Overall Study
Arm/Group | Active Comparator: Clinic Group 1 (Clinics With Existing Automated System for CSF Prescribing) | Active Comparator: Clinic Group 2 (Clinics With no Automated System for CSF Prescribing) | Experimental: Clinic Group 3 (Clinics With Automated System for CSF Prescribing) | Experimental: Clinic Group 4 (Clinics With Automated System for CSF Prescribing)
Started | 707 | 644 | 1281 | 973
Treatment Completed | 665 | 602 | 1158 | 905
Completed | 660 | 596 | 1151 | 898
Not Completed | 47 | 48 | 130 | 75
Not completed — Refusal unrelated to adverse event | 3 | 6 | 7 | 7
Not completed — Death | 44 | 42 | 123 | 68

BASELINE CHARACTERISTICS:
Groups:
- Active Comparator: Clinic Group 1 (Clinics With Existing Automated System for CSF Prescribing): CSF prescribing for patients taking anti-cancer drugs is based on existing automated system recommendations: CSF is recommended for drugs with high risk of FN; CSF is not recommended for drugs with low risk of FN.
- Active Comparator: Clinic Group 2 (Clinics With no Automated System for CSF Prescribing): CSF prescribing for patients taking anti-cancer drugs is based on existing clinical practice guidelines.
- Experimental: Clinic Group 3 (Clinics With Automated System for CSF Prescribing): CSF prescribing for patients taking anti-cancer drugs is based on automated system recommendations: CSF is recommended for drugs with intermediate or high risk of FN; CSF is not recommended for drugs with low risk of FN.
- Experimental: Clinic Group 4 (Clinics With Automated System for CSF Prescribing): CSF prescribing for patients taking anti-cancer drugs is based on automated system recommendations: CSF is recommended for drug with high risk of FN; CSF is not recommended for drugs with intermediate or low risk of FN.
- Total: Total of all reporting groups
Arm/Group | Active Comparator: Clinic Group 1 (Clinics With Existing Automated System for CSF Prescribing) | Active Comparator: Clinic Group 2 (Clinics With no Automated System for CSF Prescribing) | Experimental: Clinic Group 3 (Clinics With Automated System for CSF Prescribing) | Experimental: Clinic Group 4 (Clinics With Automated System for CSF Prescribing) | Total
Number analyzed (Participants) | 707 | 644 | 1281 | 973 | 3605
Age, Continuous [Median (Full Range); unit: years] | 58.8 [25.8 to 94.8] | 59.9 [23.6 to 86.1] | 59.6 [18.8 to 91.5] | 58.9 [22.5 to 89.7] | 59.3 [18.8 to 94.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 594 | 508 | 937 | 788 | 2827
  Male | 113 | 136 | 344 | 185 | 778
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 26 | 227 | 110 | 377
  Not Hispanic or Latino | 692 | 599 | 1012 | 846 | 3149
  Unknown or Not Reported | 1 | 19 | 42 | 17 | 79
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 22 | 17 | 40
  Asian | 10 | 15 | 45 | 24 | 94
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 7 | 6 | 14
  Black or African American | 62 | 113 | 115 | 118 | 408
  White | 622 | 500 | 1059 | 733 | 2914
  More than one race | 6 | 1 | 4 | 8 | 19
  Unknown or Not Reported | 6 | 14 | 29 | 67 | 116
Febrile Neutropenia Risk Level [Count of Participants; unit: Participants] — Febrile Neutropenia (FN) Risk Levels are defined as:
  * Low: < 10% risk of FN
  * Intermediate: 10-20% of FN
  * High: > 20% risk of FN
  Participants
    Low | 121 | 128 | 249 | 209 | 707
    Intermediate | 202 | 207 | 542 | 304 | 1255
    High | 384 | 309 | 490 | 460 | 1643
Cancer Type [Count of Participants; unit: Participants]
  Breast | 508 | 397 | 731 | 639 | 2275
  Colorectal | 136 | 181 | 368 | 245 | 930
  NSCLC | 63 | 66 | 182 | 89 | 400

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With CSF Prescribed as Primary Prophylaxis
Description: To compare the use of primary prophylactic colony stimulating factor (PP-CSF) according to recommended clinical practice guidelines among participants registered at intervention components versus usual care components. Primary prophylaxis of CSF (PP-CSF) is defined as the initiation of granulocyte CSFs during the first cycle of myelosuppressive systemic therapy, given 24 to 72 hours after cessation of systemic therapy. Separate mixed effects logistic models will be fit to assess the effect of the intervention on PP-CSF use. The rate of CSF prescribing is defined as the percent of participants prescribed CSF as primary prophylaxis out of the total number of participants within each arm.
Time Frame: Baseline to up to 14 days
Population: There was one participant in Arm 4, that was deemed as having an unavailable outcome and was excluded from this analysis population. Leaving Arm 4 with 972 analyzable participants rather than 973.
Measure: Number; unit: percentage of participants
Arm/Group | Active Comparator: Clinic Group 1 (Clinics With Existing Automated System for CSF Prescribing) | Active Comparator: Clinic Group 2 (Clinics With no Automated System for CSF Prescribing) | Experimental: Clinic Group 3 (Clinics With Automated System for CSF Prescribing) | Experimental: Clinic Group 4 (Clinics With Automated System for CSF Prescribing)
Number analyzed (Participants) | 707 | 644 | 1281 | 972
percentage of participants
  Low Risk Group: number analyzed (Participants) | 121 | 128 | 249 | 208
  Low Risk Group | 8.3 | 5.5 | 7.2 | 5.3
  Intermediate Risk Group: number analyzed (Participants) | 202 | 207 | 542 | 304
  Intermediate Risk Group | 37.1 | 18.8 | 37.1 | 9.9
  High Risk Group: number analyzed (Participants) | 384 | 309 | 490 | 460
  High Risk Group | 93.0 | 95.8 | 91.8 | 86.3
  All FN Risk Groups | 62.5 | 53.1 | 52.2 | 45.1
Statistical Analysis 1: Comparison: Active Comparator: Clinic Group 2 (Clinics With no Automated System for CSF Prescribing) vs Experimental: Clinic Group 3 (Clinics With Automated System for CSF Prescribing) vs Experimental: Clinic Group 4 (Clinics With Automated System for CSF Prescribing); PP-CSF use in the high risk FN group was compared between the usual care (UC) group (Arm 2) and the intervention group (Arm 3 and 4 combined); Test type: Superiority; p = 0.21, Regression, Logistic; Adjusted for age group, comorbidity, race, and Hispanic ethnicity; Odds Ratio (OR) = 0.44, 95% CI 2-sided [0.12 to 1.57]
Statistical Analysis 2: Comparison: Active Comparator: Clinic Group 2 (Clinics With no Automated System for CSF Prescribing) vs Experimental: Clinic Group 3 (Clinics With Automated System for CSF Prescribing) vs Experimental: Clinic Group 4 (Clinics With Automated System for CSF Prescribing); PP-CSF use in the low risk FN group was compared between the usual care (UC) group (Arm 2) and the intervention group (Arm 3 and 4 combined); Test type: Superiority; p = 0.74, Regression, Logistic; Adjusted for age, sex, and cancer type; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.44 to 3.20]
Statistical Analysis 3: Comparison: Active Comparator: Clinic Group 2 (Clinics With no Automated System for CSF Prescribing) vs Experimental: Clinic Group 3 (Clinics With Automated System for CSF Prescribing); PP-CSF use in the intermediate risk FN group was compared between the usual care (UC) group (Arm 2) and the SOE for PP-CSF intervention group (Arm 3); Test type: Superiority; p = 0.17, Regression, Logistic; Adjusted for age, sex, and cancer type; Odds Ratio (OR) = 2.23, 95% CI 2-sided [0.70 to 7.08]
Statistical Analysis 4: Comparison: Active Comparator: Clinic Group 2 (Clinics With no Automated System for CSF Prescribing) vs Experimental: Clinic Group 4 (Clinics With Automated System for CSF Prescribing); PP-CSF use in the intermediate risk FN group was compared between the usual care (UC) group (Arm 2) and the alert against PP-CSF intervention group (Arm 4); Test type: Superiority; p = 0.094, Regression, Logistic; Adjusted for age, sex, and cancer type; Odds Ratio (OR) = 0.36, 95% CI 2-sided [0.11 to 1.19]

2. Primary Outcome: Incidence of Febrile Neutropenia
Description: To compare the rate of febrile neutropenia (FN) among participants, at any risk level, registered at intervention components versus usual care components. Febrile neutropenia is defined by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0) as an absolute neutrophil count (ANC) < 1000/µL and a single temperature of > 38.3°C (101°F) or a sustained temperature of ≥ 38°C (101°F) for more than one hour.
Time Frame: Within 6 months post registration
Population: There were 18 participants deemed as having an unavailable outcome and were excluded from the analysis population, leaving 3587 analyzable participants.
Measure: Number; unit: percentage of participants
Arm/Group | Active Comparator: Clinic Group 1 (Clinics With Existing Automated System for CSF Prescribing) | Active Comparator: Clinic Group 2 (Clinics With no Automated System for CSF Prescribing) | Experimental: Clinic Group 3 (Clinics With Automated System for CSF Prescribing) | Experimental: Clinic Group 4 (Clinics With Automated System for CSF Prescribing)
Number analyzed (Participants) | 707 | 640 | 1275 | 965
percentage of participants
  Low Risk Group: number analyzed (Participants) | 121 | 127 | 245 | 207
  Low Risk Group | 1.7 | 0.8 | 1.6 | 1.5
  Intermediate Risk Group: number analyzed (Participants) | 202 | 205 | 540 | 301
  Intermediate Risk Group | 5.9 | 2.9 | 3.7 | 3.7
  High Risk Group: number analyzed (Participants) | 384 | 308 | 490 | 457
  High Risk Group | 6.5 | 4.2 | 5.7 | 6.6
  All FN Risk Groups | 5.5 | 3.1 | 4.1 | 4.6
Statistical Analysis 1: Comparison: Active Comparator: Clinic Group 2 (Clinics With no Automated System for CSF Prescribing) vs Experimental: Clinic Group 3 (Clinics With Automated System for CSF Prescribing) vs Experimental: Clinic Group 4 (Clinics With Automated System for CSF Prescribing); FN incidence rate in the high risk FN group was compared between the usual care (UC) group (Arm 2) and the intervention group (Arm 3 and 4 combined); Test type: Superiority; p = 0.26, Regression, Logistic; Adjusted for age; Odds Ratio (OR) = 1.49, 95% CI 2-sided [0.75 to 2.95]
Statistical Analysis 2: Comparison: Active Comparator: Clinic Group 2 (Clinics With no Automated System for CSF Prescribing) vs Experimental: Clinic Group 3 (Clinics With Automated System for CSF Prescribing) vs Experimental: Clinic Group 4 (Clinics With Automated System for CSF Prescribing); FN incidence rate in the low risk FN group was compared between the usual care (UC) group (Arm 2) and the intervention group (Arm 3 and 4 combined); Test type: Superiority; p = 0.51, Regression, Logistic; Adjusted for cancer type; Odds Ratio (OR) = 2.00, 95% CI 2-sided [0.23 to 18.80]
Statistical Analysis 3: Comparison: Active Comparator: Clinic Group 2 (Clinics With no Automated System for CSF Prescribing) vs Experimental: Clinic Group 3 (Clinics With Automated System for CSF Prescribing); FN incidence rate in the intermediate risk FN group was compared between the usual care (UC) group (Arm 2) and the SOE for PP-CSF intervention group (Arm 3); Test type: Superiority; p = 0.87, Regression, Logistic; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.41 to 2.88]
Statistical Analysis 4: Comparison: Active Comparator: Clinic Group 2 (Clinics With no Automated System for CSF Prescribing) vs Experimental: Clinic Group 4 (Clinics With Automated System for CSF Prescribing); FN incidence rate in the intermediate risk FN group was compared between the usual care (UC) group (Arm 2) and the alert against PP-CSF intervention group (Arm 4); Test type: Superiority; p = 0.68, Regression, Logistic; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.44 to 3.57]

3. Primary Outcome: Incidence of Febrile Neutropenia Among Intermediate Risk Participants
Description: To compare the rate of FN among intermediate risk participants registered at intervention components by component treatment assignment (administer PP-CSF to intermediate risk participants versus not). Febrile neutropenia is defined by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0) as an absolute neutrophil count (ANC) < 1000/µL and a single temperature of > 38.3°C (101°F) or a sustained temperature of ≥ 38°C (101°F) for more than one hour.
Time Frame: Within 6 months post registration
Population: The analysis population includes only participants that are classified as having intermediate risk of FN. Seven participants were deemed as having an unavailable outcome and were excluded from the analysis population.
Measure: Number; unit: percentage of participants
Arm/Group | Active Comparator: Clinic Group 1 (Clinics With Existing Automated System for CSF Prescribing) | Active Comparator: Clinic Group 2 (Clinics With no Automated System for CSF Prescribing) | Experimental: Clinic Group 3 (Clinics With Automated System for CSF Prescribing) | Experimental: Clinic Group 4 (Clinics With Automated System for CSF Prescribing)
Number analyzed (Participants) | 202 | 205 | 540 | 301
percentage of participants | 5.9 | 2.9 | 3.7 | 3.7
Statistical Analysis 1: Comparison: Experimental: Clinic Group 3 (Clinics With Automated System for CSF Prescribing) vs Experimental: Clinic Group 4 (Clinics With Automated System for CSF Prescribing); Test type: Superiority; p = 0.74, Regression, Logistic; Adjusted for cancer type; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.39 to 1.95]
Statistical Analysis 2: Comparison: Active Comparator: Clinic Group 2 (Clinics With no Automated System for CSF Prescribing) vs Experimental: Clinic Group 3 (Clinics With Automated System for CSF Prescribing); Test type: Superiority; p = 0.87, Regression, Logistic; Adjusted for cancer type; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.41 to 2.88]
Statistical Analysis 3: Comparison: Active Comparator: Clinic Group 2 (Clinics With no Automated System for CSF Prescribing) vs Experimental: Clinic Group 4 (Clinics With Automated System for CSF Prescribing); This is comparing the FN incidence rate in the arm randomized to alert against PP-CSF vs usual care in intermediate risk participants; Test type: Superiority; p = 0.68, Regression, Logistic; Adjusted for cancer type; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.44 to 3.57]

4. Secondary Outcome: Incidence of Febrile Neutropenia Among Low Risk Participants
Description: To compare the rate of FN among low-risk participants registered at intervention components versus usual care components. Febrile neutropenia is defined by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0) as an absolute neutrophil count (ANC) < 1000/µL and a single temperature of > 38.3°C (101°F) or a sustained temperature of ≥ 38°C (101°F) for more than one hour.
Time Frame: Within 6 months of registration
Population: The analysis population includes only participants deemed 'low-risk' within each of the clinic groups.
Measure: Number; unit: percentage of participants
Arm/Group | Active Comparator: Clinic Group 1 (Clinics With Existing Automated System for CSF Prescribing) | Active Comparator: Clinic Group 2 (Clinics With no Automated System for CSF Prescribing) | Experimental: Clinic Group 3 (Clinics With Automated System for CSF Prescribing) | Experimental: Clinic Group 4 (Clinics With Automated System for CSF Prescribing)
Number analyzed (Participants) | 111 | 120 | 229 | 196
percentage of participants | 1.8 | 0.8 | 1.8 | 1.5

5. Secondary Outcome: FN-related Health-Related Quality of Life (HRQOL) Among Low Risk Participants
Description: To compare the FN-related health-related quality of life (HRQOL) among low-risk participants registered at intervention components versus usual care components. Assessed using the Functional Assessment of Cancer Therapy - Febrile Neutropenia (Version 4) (FACT-N). Includes FACT general cancer score and FN-related score. A linear mixed effects model will be fit to assess the effect of the intervention on HRQOL. Component-level characteristics, patient-level clinical and demographic variables will be adjusted.
Time Frame: Baseline to up to 14 days
Reporting Status: Not Posted

6. Secondary Outcome: Participant Adherence Rates to PP-CSF Prescription
Description: To compare adherence to PP-CSF prescribing among participants registered at intervention components versus usual care components. Participant adherence rates are obtained from the proportion receiving PP-CSF among those for whom PP-CSF was ordered by the physician. The primary adherence measure will be obtained from the participant's chart; secondary adherence will be measured via self-report on the Follow-Up Participant Survey. For the home and clinic settings, separate mixed effects logistic models will be used to assess the effect of the intervention on adherence to PP-CSF orders, treating adherence after the start of the study. Component-level characteristics, participant-level clinical and demographic variables will be adjusted.
Time Frame: Within 14 days after the completion of first course of therapy
Reporting Status: Not Posted

7. Secondary Outcome: Change in Participant Knowledge of PP-CSF Indications
Description: To compare participant knowledge of the indications for, efficacy of, and side effects associated with PP-CSF between the initiation and conclusion of the first cycle of myelosuppressive systemic therapy among participants registered at intervention components versus usual care components. Linear mixed effects model with a time variable and an interaction between randomized group and time will be used to analyze change in the patient knowledge score. Random effects will be used to accommodate both the correlation among measures from the same patient as well as the correlation among patients from the same component. Component-level characteristics, participant-level clinical and demographic variables will be adjusted.
Time Frame: Baseline to up to 14 days
Reporting Status: Not Posted

8. Secondary Outcome: Proportion Completing Initial Systemic Therapy Regimen: a) at Planned Duration and b) at Planned Dose Intensity (Clinical)
Description: To compare the proportion of participants completing the initial systemic therapy regimen at planned duration and at planned dose intensity among participants registered at intervention components versus usual care components.Two separate mixed effects logistic models will be used to assess the effect of the intervention on completion of the initial systemic therapy regimen (i) at planned duration and (ii) at planned dose intensity. Component-level characteristics, patient-level clinical and demographic variables will be adjusted.
Time Frame: Up to 12 months
Reporting Status: Not Posted

9. Secondary Outcome: Prophylactic and FN-Related Antibiotic Use
Description: To compare antibiotic use both as prophylaxis and as treatment for FN among participants registered at intervention components versus usual care components. Prophylactic and FN-related antibiotic use will be measured as total number of antibiotic agents used and duration of antibiotic use. A linear mixed effects model will be fit to assess the effect of the intervention on duration of antibiotics use with number of days. Mixed effects Poisson models will be used to assess the effect of the intervention on total number of antibiotics agents used. Three separate models will be fit, with the following outcomes: (i) the number of times antibiotics were used as prophylaxis, (ii) the number of times antibiotics were used as treatment for FN, and (iii) t
Time Frame: Within 30 days of therapy
Reporting Status: Not Posted

10. Secondary Outcome: Rate of FN-Related Emergency Department Visits and Hospitalizations
Description: To compare the rate of FN-related emergency department (ED) visits and hospitalizations among intermediate risk participants registered to intervention components by component treatment assignment (administer PP-CSF to intermediate risk participants versus not). FN-related ED visits and hospitalizations are defined as admission to ED or hospital with documentation of fever and decreased ANC. A mixed effects Poisson model will be used to assess the effect of the intervention on FN-related ED visits and hospitalizations. Robust variance estimation will be used to relax the strong assumptions about the variance made by Poisson regression. If a large number of zero counts is observed, then zero-inflated Poisson regression will be used.
Time Frame: At 6 months
Reporting Status: Not Posted

11. Secondary Outcome: FN-related Health-Related Quality of Life (HRQOL) Among Intermediate Risk Participants
Description: To compare the FN-related health-related quality of life (HRQOL) among intermediate risk participants registered to intervention components by component treatment assignment (administer PP-CSF to intermediate risk participants versus not). Assessed using the Functional Assessment of Cancer Therapy - Febrile Neutropenia (Version 4) (FACT-N). Includes FACT general cancer score and FN-related score. A linear mixed effects model will be fit to assess the effect of the intervention on HRQOL. Component-level characteristics, participant-level clinical and demographic variables will be adjusted.
Time Frame: Baseline to up to 14 days
Reporting Status: Not Posted

12. Secondary Outcome: Overall Survival (OS)
Description: To compare overall survival among intermediate risk participants registered to intervention components by component treatment assignment (administer PP-CSF to intermediate risk participants versus not). A Cox proportional hazards model will be used to model survival. Component-level characteristics, participant-level clinical and demographic variables will be adjusted. A separate analysis of cause-specific survival to address FN-related deaths will also be conducted.
Time Frame: Time from date of registration to date of death due to any cause, assessed up to 12 months
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Time to Invasive Recurrence in Non-Metastatic Participants
Description: To evaluate the time to invasive recurrence in non-metastatic participants by component treatment assignment. Analysis will be exploratory and comparative.
Time Frame: Time from registration to documented invasive local or regional recurrence, assessed up to 12 months
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Differences Among Cohort Components and Intervention and Usual Care Components
Description: To characterize and descriptively report the differences among cohort components and the intervention and usual care components.
Time Frame: Up to 12 months post registration
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were monitored/assessed through the end of first anti-cancer treatment cycle, an average of 21 days. While All-Cause Mortality was monitored/assessed for the entire duration participants are followed for the study, an average of 12 months.
Description: Adverse events (AEs) are reported by CTCAE version 4.0. Only participants that received PP-CSF during the first cycle of anti-cancer treatment were evaluated for adverse events. Population at risk for all-cause mortality includes all eligible and analyzable participants regardless of if they received PP-CSF.
Arm/Group | Active Comparator: Clinic Group 1 (Clinics With Existing Automated System for CSF Prescribing) | Active Comparator: Clinic Group 2 (Clinics With no Automated System for CSF Prescribing) | Experimental: Clinic Group 3 (Clinics With Automated System for CSF Prescribing) | Experimental: Clinic Group 4 (Clinics With Automated System for CSF Prescribing)
All-Cause Mortality (participants affected / at risk) | 44/707 | 42/644 | 123/1281 | 68/973
Serious Adverse Events (participants affected / at risk) | 3/456 | 0/350 | 0/694 | 1/448
Other Adverse Events (participants affected / at risk) | 146/456 | 123/350 | 243/694 | 171/448
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Comparator: Clinic Group 1 (Clinics With Existing Automated System for CSF Prescribing) (N=456) | Active Comparator: Clinic Group 2 (Clinics With no Automated System for CSF Prescribing) (N=350) | Experimental: Clinic Group 3 (Clinics With Automated System for CSF Prescribing) (N=694) | Experimental: Clinic Group 4 (Clinics With Automated System for CSF Prescribing) (N=448)
Sepsis (Infections and infestations) | 1 | 0 | 0 | 1
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active Comparator: Clinic Group 1 (Clinics With Existing Automated System for CSF Prescribing) (N=456) | Active Comparator: Clinic Group 2 (Clinics With no Automated System for CSF Prescribing) (N=350) | Experimental: Clinic Group 3 (Clinics With Automated System for CSF Prescribing) (N=694) | Experimental: Clinic Group 4 (Clinics With Automated System for CSF Prescribing) (N=448)
Mucositis oral (Gastrointestinal disorders) | 10 | 13 | 44 | 27
Arthralgia (Musculoskeletal and connective tissue disorders) | 51 | 44 | 81 | 76
Bone pain (Musculoskeletal and connective tissue disorders) | 110 | 101 | 205 | 121
Myositis (Musculoskeletal and connective tissue disorders) | 6 | 2 | 24 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-11-13): https://cdn.clinicaltrials.gov/large-docs/96/NCT02728596/Prot_SAP_ICF_000.pdf